CLINICAL TRIAL: NCT07111520
Title: A Phase Ib/II, Multi-site, Open-label, Dose Finding Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of BNT326 in Combination With BNT327 in Participants With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Clinical Trial to Test if an Investigational Combination Therapy With BNT326 and BNT327 is Safe and Potentially Beneficial for People With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT326-02; 2024-519344-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Combination with other investigational agents; Programmed death-ligand 1 (PD-L1); Antibody-drug conjugate (ADC); Human epidermal growth factor receptor 3 (HER3); Programmed Death-1 (PD-1); Programmed Death-1 monoclonal antibodies; Combination chemotherapy; Anti vascular endothelial growth factor-A (anti-VEGF-A); Bispecific antibody; Immunotherapy; Dose optimization; Time to progression; Vascular endothelial growth factor (VEGF)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lethal Congenital Contracture Syndrome 2 | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part 1 - BNT326 (DL1, starting dose) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with second-line (or higher) 2L(+), squamous or non-squamous NSCLC, actionable genomic alterations (AGA)-negative/positive, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 1 - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L(+), squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 1 - BNT326 (DL3, optional) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L(+), squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2a (Cohort A, Arm 1) - BNT326 (DL1) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L+ squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2a (Cohort A, Arm 2) - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L+ squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2a (Cohort B, Arm 1) - BNT326 (DL1) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with first-line (1L) squamous or non-squamous NSCLC, AGA-negative, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2a (Cohort B, Arm 2) - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 1L squamous or non-squamous NSCLC, AGA-negative, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2b (Cohort C, Arm 1) - BNT326 (DL1) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L+, squamous or non-squamous NSCLC, AGA-negative or epithelial growth factor receptor (EGFR) activating mutation, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2b (Cohort C, Arm 2) - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 2L+, squamous or non-squamous NSCLC, AGA-negative or EGFR activating mutation, any PD-L1.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2b (Cohort C, Arm 3) - BNT326 monotherapy (Experimental): BNT326 monotherapy (DL2). In participants with 2L+, squamous or non-squamous NSCLC, AGA-negative or EGFR activating mutation, any PD-L1.
  Interventions: Drug: BNT326
- Part 2b (Cohort D1, Arm 1) - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 ≥50%.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2b (Cohort D1, Arm 2) - Pembrolizumab (Active Comparator): Pembrolizumab monotherapy. In participants with 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 ≥50%.
  Interventions: Drug: Pembrolizumab
- Part 2b (Cohort D1, Arm 3) - BNT327 monotherapy (Experimental): BNT327 monotherapy. In participants with 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 ≥50%.
  Interventions: Drug: BNT327
- Part 2b (Cohort D2, Arm 1) - BNT326 (DL2) + BNT327 (Experimental): Combination therapy of BNT326 and BNT327. In participants with 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 <50%.
  Interventions: Drug: BNT326; Drug: BNT327
- Part 2b (Cohort D2, Arm 2) - SoC - Pembrolizumab + chemotherapy (Active Comparator): Combination therapy of pembrolizumab and chemotherapy. In participants with 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 <50%.
  Interventions: Drug: Pembrolizumab; Drug: SoC

INTERVENTIONS:
Drug: BNT326 — intravenous (IV) infusion
  Arms: Part 1 - BNT326 (DL1, starting dose) + BNT327; Part 1 - BNT326 (DL2) + BNT327; Part 1 - BNT326 (DL3, optional) + BNT327; Part 2a (Cohort A, Arm 1) - BNT326 (DL1) + BNT327; Part 2a (Cohort A, Arm 2) - BNT326 (DL2) + BNT327; Part 2a (Cohort B, Arm 1) - BNT326 (DL1) + BNT327; Part 2a (Cohort B, Arm 2) - BNT326 (DL2) + BNT327; Part 2b (Cohort C, Arm 1) - BNT326 (DL1) + BNT327; Part 2b (Cohort C, Arm 2) - BNT326 (DL2) + BNT327; Part 2b (Cohort C, Arm 3) - BNT326 monotherapy; Part 2b (Cohort D1, Arm 1) - BNT326 (DL2) + BNT327; Part 2b (Cohort D2, Arm 1) - BNT326 (DL2) + BNT327
Drug: BNT327 — IV infusion
  Arms: Part 1 - BNT326 (DL1, starting dose) + BNT327; Part 1 - BNT326 (DL2) + BNT327; Part 1 - BNT326 (DL3, optional) + BNT327; Part 2a (Cohort A, Arm 1) - BNT326 (DL1) + BNT327; Part 2a (Cohort A, Arm 2) - BNT326 (DL2) + BNT327; Part 2a (Cohort B, Arm 1) - BNT326 (DL1) + BNT327; Part 2a (Cohort B, Arm 2) - BNT326 (DL2) + BNT327; Part 2b (Cohort C, Arm 1) - BNT326 (DL1) + BNT327; Part 2b (Cohort C, Arm 2) - BNT326 (DL2) + BNT327; Part 2b (Cohort D1, Arm 1) - BNT326 (DL2) + BNT327; Part 2b (Cohort D1, Arm 3) - BNT327 monotherapy; Part 2b (Cohort D2, Arm 1) - BNT326 (DL2) + BNT327
Drug: Pembrolizumab — IV infusion
  Arms: Part 2b (Cohort D1, Arm 2) - Pembrolizumab; Part 2b (Cohort D2, Arm 2) - SoC - Pembrolizumab + chemotherapy
Drug: SoC — IV infusion. Combination chemotherapy (pemetrexed, paclitaxel, or carboplatin). Chemotherapy will be selected according to the indication.
  Arms: Part 2b (Cohort D2, Arm 2) - SoC - Pembrolizumab + chemotherapy

SUMMARY:
This is a multi-site, open-label, dose-finding study, consisting of Parts 1, 2a, and 2b to investigate the combination of BNT326 with BNT327 in participants with relapsed, progressive as well as treatment-naïve, advanced/metastatic non-small cell lung cancer (NSCLC).

This study will enroll adult participants with histologically or cytologically confirmed NSCLC that is advanced (i.e., either metastatic or recurrent tumors with no known curative treatment available).

DETAILED DESCRIPTION:
Part 1 is a dose escalation to evaluate and establish two or three safe combination dose levels (DL1 and DL2 and optionally DL3) of BNT326 with BNT327.

Part 2a is a dose expansion to evaluate the preliminary efficacy, safety, and tolerability.

Part 2b is a dose optimization and contribution of components part.

Parts 1 and 2a (Cohort A) will enroll participants with previous exposure to therapy for advanced/metastatic disease. Part 2a (Cohort B) and Part 2b (Cohorts C and D) will enroll less heavily pre-treated participants, namely those without prior systemic treatment for advanced/metastatic disease.

The sponsor, having heard the internal review committee, may determine the dose levels for each arm in Cohorts C and D based on data generated from Parts 1 and 2a. The dose levels chosen for Cohorts C and D will not exceed the highest dose level investigated in this study.

Parts 1 and 2a will be non-randomized. In Part 2b, participants will be randomized to different treatments within each cohort.

The study consists of a screening period, a treatment period, a safety follow-up period, an efficacy follow-up period, and a long-term survival follow-up. Participants will receive study treatment until disease progression, withdrawal of consent, termination of the study by the sponsor, unacceptable toxicity, or for a maximum duration of 24 months (or for the maximum duration as per the local product label for participants receiving standard of care [SoC] therapy), whichever occurs first. For each study participant, the treatment and follow-up periods are projected to be completed within ~36 months, unless participants are continuing to benefit from treatment per investigator's recommendation and upon sponsor approval.

ELIGIBILITY:
Key Inclusion Criteria (applicable to all participants and all parts unless otherwise specified):

* Aged ≥18 years at the time of giving informed consent.
* Have measurable disease defined by RECIST v1.1.
* All participants have to provide a tumor tissue sample (e.g. Formalin-fixed paraffin-embedded [FFPE] slides or block) from archival tissue. Alternatively, a fresh biopsy should be collected, unless medically not justifiable to be conducted.
* Have Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have adequate organ and bone marrow function within 7 days before randomization/enrollment.
* Have advanced (i.e., metastatic or locally recurrent where local therapy with curative intent is not possible) non-squamous or squamous (all cohorts) or only non-squamous (Cohort D2) NSCLC.

Cohort-specific inclusion criteria

Part 1, 2L+, squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1

* for AGA-negative NSCLC only:

  * Have no actionable genomic alterations, such as EGFR mutations, anaplastic lymphoma kinase (ALK) gene rearrangements, or other genomic alterations for which targeted molecular therapies are available.
  * Have experienced relapse or progression during or after treatment with standard systemic therapy in the advanced/metastatic setting or discontinued from prior therapy due to intolerance.
  * Participants must have received 1 to 3 lines of systemic treatment, which can include anti-PD-1/PD-L1 therapy, chemotherapy, and anti-angiogenic agents. These treatments may be administered concurrently or sequentially. However, chemotherapy treatment must be limited to 2 lines or less.
* for AGA-positive NSCLC only (excluding EGFR activating mutation):

  * Have documented positive test results for one or more actionable genomic alteration: EGFR (other than activating mutations), ALK, ROS proto-oncogene 1 (ROS1), gene encoding the hepatocyte growth factor receptor (MET), human gene that encodes a protein called B-Raf (BRAF), rearranged during transfection (RET), neurotrophic tropomyosin-receptor kinase (NTRK), human epidermal growth factor receptor 2 (HER2), Kirsten rat sarcoma virus (KRAS), or other genomic alteration with available targeted therapy.
  * Must have received at least one prior systemic therapy for advanced disease, which must have included targeted treatment for actionable genomic alterations, which include alterations such as EGFR (other than activating mutations), ALK, ROS1, MET, BRAF, RET, NTRK, HER2, KRAS, or other alterations for which targeted therapies are available as a part of local SoC.
  * Participants may have received between 1 to 3 lines of systemic treatment of anti-PD-1/PD-L1 therapy, chemotherapy, and/or anti-angiogenic agents. These treatments may be administered concurrently (including with TKI) or sequentially. However, chemotherapy treatment must be limited to 2 lines or less.
  * Have experienced progression during or after treatment or discontinued from prior therapy due to intolerance.
* for AGA-positive NSCLC only (with EGFR activating mutation):

  * Have documented positive test results for an EGFR-sensitizing mutation (EGFR-sensitizing mutation Exon 21-L858R and 19del).
  * Participants must have received one or two prior lines of systemic therapy for advanced and/or metastatic disease, which must include treatment with an approved EGFR TKI, with at least one being a third-generation EGFR TKI.
  * Participants receiving an EGFR TKI at the time of signing informed consent may continue to take the EGFR TKI until 5 days prior to Cycle 1 Day 1.
  * Chemotherapy is permitted only if it was administered in combination with an EGFR TKI as part of a single line of therapy and as the initial (first line) treatment for advanced/metastatic disease.
  * Have experienced progression during or after treatment or discontinued from prior therapy due to intolerance.

Part 2a (Cohort A), 2L+, squamous or non-squamous NSCLC, AGA-negative/positive, any PD-L1

* for AGA-positive NSCLC only, excluding EGFR activating mutation:

  * Have documented positive test results for one or more actionable genomic alterations: EGFR (other than activating mutations), ALK, ROS1, MET, BRAF, RET, NTRK, HER2, KRAS, or other genomic alterations, with available targeted therapy.
  * May have received 1 to 4 lines of systemic treatment, of which one prior systemic therapy for advanced disease must have included targeted treatment for actionable genomic alterations, which include alterations such as EGFR (other than activating mutations), ALK, ROS1, MET, BRAF, RET, NTRK, HER2, KRAS, or other genomic alterations for which targeted therapies are available as part of local SoC.
  * Other therapies may include anti-PD-1/PD-L1 therapy, chemotherapy, and anti-angiogenic agents. These treatments may be administered concurrently/in combination (including with TKI) or sequentially. However, chemotherapy treatment must be limited to 2 lines or less.
  * Have experienced progression during or after treatment or discontinued from prior therapy due to intolerance.
* for AGA-positive NSCLC only, with EGFR activation mutation:

  * Have documented positive test results for an EGFR-sensitizing mutation (EGFR-sensitizing mutation Exon 21-L858R and 19del).
  * Participants must have received one or two prior lines of systemic therapy for advanced and/or metastatic disease, which must include treatment with an approved EGFR TKI, with at least one being a third-generation EGFR TKI.
  * Participants receiving an EGFR TKI at the time of signing informed consent may continue to take the EGFR TKI until 5 days prior to Cycle 1 Day 1.
  * Chemotherapy is permitted only if it was administered in combination with an EGFR TKI as part of a single line of therapy and as the initial (first line) treatment for advanced/metastatic disease.
  * Have experienced progression during or after treatment or discontinued from prior therapy due to intolerance.

Part 2a (Cohort B), 1L, squamous or non-squamous NSCLC, AGA-negative, any PD-L1

* Have no actionable genomic alterations, such as EGFR mutations, ALK rearrangements, or other genomic alterations for which targeted molecular therapies are available.
* Have received no systemic anti-cancer treatment in the advanced/metastatic setting. May have received neoadjuvant and/or adjuvant treatment if progression to advanced/metastatic disease occurred at least 12 months after completing such therapy and have not received treatment in the advanced/metastatic setting.

Part 2b (Cohort C), 2L+, squamous or non-squamous NSCLC, AGA-negative or EGFR activating mutation, any PD-L1

* for AGA-negative NSCLC only:

  * Have no actionable genomic alterations, such as EGFR mutations, ALK rearrangements, or other genomic alterations for which targeted molecular therapies are available.
  * Participants should have received 1 to 4 lines of systemic treatment, which can include anti-PD-1/PD-L1 therapy, chemotherapy, and/or anti-angiogenic agents.
* for EGFR-sensitizing mutation NSCLC only:

  * Have documented positive test results for an EGFR-sensitizing mutation (EGFR-sensitizing mutation Exon 21-L858R and 19del).
  * Have received 1 or 2 prior systemic therapies for advanced and/or metastatic disease with an approved EGFR TKI, which must include one third-generation anti-EGFR TKI.
  * Participants receiving an EGFR TKI at the time of signing informed consent may continue to take the EGFR TKI until 5 days prior to Cycle 1 Day 1.
  * Chemotherapy is permitted only if it was administered in combination with an EGFR TKI as part of a single line of therapy and as the initial (first line) treatment for advanced/metastatic disease.
  * May have received neoadjuvant and/or adjuvant treatment if progression to advanced/metastatic disease occurred at least 6 months after completing such therapy and have experienced disease progression on or after EGFR TKI treatment administered in the advanced/metastatic setting.
  * Have experienced progression during or after treatment or discontinued from prior therapy due to intolerance.

Part 2b (Cohort D1) 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 ≥50% and Part 2b (Cohort D2) 1L, squamous or non-squamous NSCLC, AGA-negative, PD-L1 <50%

* Have no actionable genomic alterations, such as EGFR mutations, ALK rearrangements, or other genomic alterations for which targeted molecular therapies are available.
* Did not receive prior systemic therapy for advanced and/or metastatic disease.

Key Exclusion Criteria (applicable to all participants and all parts):

* Had disease progression on or were intolerant to prior treatment with an agent targeting HER3 (including antibody, ADC, cell therapy, and other drugs) or with a topoisomerase I inhibitor payload (including topoisomerase I inhibitor-containing ADCs). Note: For Part 2a Cohort A, prior exposure to agents targeting HER3 or topoisomerase I inhibitor payload may be allowed on a case-by-case basis after discussion with and approval by the sponsor.
* Have an uncontrolled concomitant or intercurrent illness, that contra-indicates study participation, limits compliance with study procedures or substantially increases the risk of incurring AEs, including:

  * Bleeding diathesis or active hemorrhage
  * Active infection, including respiratory viral infection
  * Child-Pugh class B or C cirrhosis
  * Known pulmonary disease with significant impact in lung function and/or with potential risk of severe infection
  * Oncologic emergencies or complications (e.g., malignant hypercalcemia, superior vena cava syndrome, carcinoid syndrome that is unstable and with available alternative therapies)
  * Psychiatric or abuse condition
  * Colitis Grade ≥2 not resolved within 72 h within the past 3 months
* Have left ventricular ejection fraction <50% by either echocardiography or multi-gated acquisition (scanning) within 28 days before randomization/enrollment.
* Have clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy within 2 weeks prior to randomization/enrollment.
* Have a history of (non-infectious) interstitial lung disease (ILD) /pneumonitis that required steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening. Asymptomatic interstitial changes caused by previous radiation therapy, chemotherapy, or other factors such as smoking are acceptable.
* Have had exposure to protocol-specific treatments with a washout period before randomization/enrollment.
* Are participants of childbearing potential who are pregnant or breastfeeding or are planning pregnancy within the time specified in the protocol or are potentially fertile males, who are planning to father children during the study or within the time specified in the protocol.
* Are subject to exclusion periods from another investigational study.
* Have a history of small bowel obstruction requiring hospitalization within the past 3 months prior to the first dose of IMP.
* Have urine protein ≥2+ and 24-hour urine protein excretion ≥1 g. If qualitative urine protein is ≤1+, a 24-hour urine protein quantitative test is not required.
* Have a history of Grade ≥3 immune-related adverse events that led to treatment discontinuation of a prior checkpoint inhibitor.
* Have clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Participants with significant risks of hemorrhage or evidence of major coagulation disorders.
* Have active or chronic corneal disorders or with any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Occurrence of dose limiting toxicities (DLTs) within a participant | 21 days starting on Day 1 of Cycle 1
  During the DLT evaluation period by dose level
Part 1 and Part 2a - Occurrence of treatment emergent adverse events (TEAEs), treatment-related adverse events (TRAE), treatment emergent serious adverse events (TESAE), treatment-related serious adverse events (TRSAE) | from the first dose of investigational medicinal product (IMP) up to 90 days after the last dose of IMP or until a new systemic anti-cancer therapy is started, whichever occurs first (up to a maximum of 27 months)
Part 1 and Part 2a - Occurrence of dose interruption, reduction, and discontinuation due to TEAEs | from the first dose of IMP up to 90 days after the last dose of IMP or until a new systemic anti-cancer therapy is started, whichever occurs first (up to a maximum of 27 months)
Part 2a and Part 2b - Objective response rate (ORR) | from the time of initiation of the first dose of IMP to approximately 36 months
  Defined as the percentage of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] based on the investigator's assessment) is observed as best overall response.

SECONDARY OUTCOMES:
Part 1 - ORR | from the time of initiation of the first dose of IMP to approximately 36 months
  Defined as the percentage of participants in whom a confirmed CR or PR (per RECIST v1.1 based on the investigator's assessment) is observed as best overall response.
Part 2b - Occurrence of TEAEs, TRAEs, TESAEs, TRSAEs | from the first dose of IMP up to 90 days after the last dose of IMP or until a new systemic anti-cancer therapy is started, whichever occurs first (up to a maximum of 27 months)
Part 2b - Occurrence of dose interruption, reduction, and discontinuation due to TEAEs | from the first dose of IMP up to 90 days after the last dose of IMP or until a new systemic anti-cancer therapy is started, whichever occurs first (up to a maximum of 27 months)
Part 2a and Part 2b - Progression free survival based on the investigator's assessment | from the first dose of IMP to approximately 36 months
  Defined as the time from first dose of IMP to the first objective tumor progression (progressive disease [PD] per RECIST v1.1) or death from any cause, whichever occurs first.
Part 2a and Part 2b - Disease control rate | from the first dose of IMP to approximately 36 months
  Defined as the proportion of participants with CR, PR, or stable disease (per RECIST v1.1 based on the investigator's assessment) as best overall response.
Part 2a and Part 2b - Duration of response | from the first dose of IMP to approximately 36 months
  Defined as the time from first confirmed objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) to first occurrence of objective tumor progression (PD per RECIST v1.1 based on the investigator's assessment) or death from any cause, whichever occurs first
Part 2a and Part 2b - Time to response | from the first dose of IMP to approximately 36 months
  Defined as the time from first dose of IMP to first confirmed objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) in participants with a confirmed objective response
Part 2a and Part 2b - Overall survival | from the first dose of IMP to approximately 36 months
  Defined as the time from first dose of IMP to death from any cause
All cohorts - PK assessment: Maximum concentration derived from serum concentrations of BNT326 ADC, total anti-HER3 antibody component, and unconjugated payload | from the first IMP up to safety follow-up, approximately 90 days post last IMP dose
  For applicable participants, if data permits.
All cohorts - PK assessment: Time to reach maximum (peak) serum concentration derived from serum concentrations of BNT326 ADC, total anti-HER3 antibody component, and unconjugated payload | from the first dose of IMP up to safety follow-up, approximately 90 days post last IMP dose
  For applicable participants, if data permits.
All cohorts - Anti-drug antibody (ADA) prevalence and ADA incidence | up to 1 year from the last dose of IMP
  By cohort and combination treatment regimen for applicable participants

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (2):
- NEXT Virginia, Fairfax, Virginia, United States
- Institute of Oncology, ARENSIA Exploratory Medicine, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No